CLINICAL TRIAL: NCT01545206
Title: Better Quality With Less Cost? A Single Hospital Experience on Reducing Door-to-balloon Time in ST-elevation Myocardial Infarction
Brief Title: Dose Reducing Door-to-balloon Time in ST-elevation Myocardial Infarction Cause Less Cost?
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chieh-Min Fan, Attending Physician, Far Eastern Memorial Hospital
Other Study IDs: 100046-E
Record Dates: First submitted 2012-03-01; First posted 2012-03-06 (Estimated); Last update posted 2012-03-06 (Estimated); Status verified 2012-03

CONDITIONS: Acute STEMI; Primary Percutaneous Coronary Arterial Intervention
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- acute STEMI, Primpary PCI

SUMMARY:
The investigators tried to determined whether the less D2B time led to costs savings benefited insurance payer and better outcomes to patients.

DETAILED DESCRIPTION:
The relationship between the quality of care and costs has been discussed widely. Higher costs of care did not bring better outcomes, vice versa. However, as the rising spending of health care, the health care providers, insurance payers, governments, and consumers begin to pursue the higher quality of cares with lowest costs. In surgical experiences, improving the process of care succeeded to improve the quality of care and reduce the costs.

In patients with acute ST-Segment elevation myocardial infarction (STEMI), A Door-to-Balloon (D2B) time of less than 90 minutes has been established as the gold standard for primary percutaneous coronary intervention (PCI) and was associated with lower in-hospital mortality.9 Only less literatures discussed the costs and the quality of care in acute STEMI, and whether improving processes of care associated with lower costs was still controversial. The Premier Hospital Quality Incentive Demonstration (PHQID) in United State improved the processes of care but had not a significant effect on cost. Another single hospital experience in Indiana, USA, showed that the reducing D2B time in STEMI decreased the insurance payments as well as the total hospital costs. However, this study design was before-and-after intervention analysis, did not actually measure the impact of D2B time. Besides, the payment system in this study was prospective payment, not fee-for-service payment in Taiwan.

In this study, we tried to determined whether the less D2B time led to costs savings benefited insurance payer and better outcomes to patients.

ELIGIBILITY:
Inclusion Criteria:

* self visit
* acute STEMI by ECG definition

Exclusion Criteria:

* non-diagnosis on first ECG
* transferred
* diagnostic angiogram only

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient presented between Feb. 1, 2007 and Jul. 31, 2009 at Far Eastern Memory Hospital for acute STEMI and unwent primary PCI.
Sampling Method: Non-Probability Sample
Enrollment: 215 (Actual)
Dates: Start 1997-02; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chieh-Min Fan, MD, MSc, Principal Investigator — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, Taipei, Taiwan